CLINICAL TRIAL: NCT02080962
Title: Hypofractionated Radiotherapy for Nonmelanoma Skin Cancer: Study Phase II Clinical Trial
Brief Title: Hypofractionated Radiotherapy for Nonmelanoma Skin Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low rate of recruitment.
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 399/2010
Record Dates: First submitted 2014-02-03; First posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Non-melanoma Skin Cancer
Keywords: non-melanoma skin cancer, radiotherapy, orthovoltage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 Gy in 5 fractions of 6 Gy (Experimental): tumors ≤ 2 cm in diameter: 5 fractions of 600 cGy, once a day, five times a week - TDF: 89
  Interventions: Radiation: 30 Gy in 5 fractions
- 40 Gy in 10 fractions of 4 Gy (Experimental): tumors > 2-5 cm in diameter: 10 fractions of 400 cGy, once a day, five times a week - TDF: 96
  Interventions: Radiation: 40 Gy in 10 fractions

INTERVENTIONS:
Radiation: 30 Gy in 5 fractions — 5 fractions of 600 cGy, once a day, five times a week - TDF: 89
  Other Names: hypofractionated orthovoltage
  Arms: 30 Gy in 5 fractions of 6 Gy
Radiation: 40 Gy in 10 fractions — tumors > 2-5 cm in diameter: 10 fractions of 400 cGy, once a day, five times a week - TDF: 96
  Other Names: hypofractionated orthovoltage
  Arms: 40 Gy in 10 fractions of 4 Gy

SUMMARY:
Radiotherapy is a treatment considered standard for non melanoma skin cancer. This institution uses schemes of 4 to 6 weeks of treatment. The objective of the study is to perform radiation therapy in 1 to 2 weeks, depending on the size of the lesion.

DETAILED DESCRIPTION:
Delineation of radiation field

* Gross tumor volume (GTV): disease clinically visible / palpable
* clinical target volume (CTV): equal to GTV
* planned treatment volume (PTV):
* tumors ≤ 2 cm in diameter, with 5-10 mm CTV margin
* tumors> 2-5 cm in diameter, with 15-20 mm CTV margin
* Marking the GTV and PTV pen back projection
* photograph of the treatment area
* protections of the normal structures with blocks of lead, if necessary

Technical

* Distance focus-skin Tube: 35 cm Locator: 30 and 40 cm
* Sizes Tube: 2, 3 and 4 cm in diameter Finder: 6x8 cm, 8x10 cm
* Energy:

  80 kV 140 kv
* Filter 80 kV, 2 mm Al 140 kv, 0.5 mm Copper
* Current Draw: 20 mA

Dose

* tumors ≤ 2 cm in diameter: 5 fractions of 600 cGy, once a day, five times a week - TDF: 89
* tumors > 2-5 cm in diameter: 10 fractions of 400 cGy, once a day, five times a week - TDF: 96

Clinical revisions every 5 weekly sessions, or a weekly and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cosmesis not important
* Basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) of any differentiation
* Clinical stage I and II
* Location on the thorax, abdomen, pelvis (except perineum), arm, thigh, cheek
* Patient with up to 3 injuries eligible for the study
* Karnofsky Performance Status (KPS) ≥ 70%
* Age > 18 years
* Informed Consent signed by the patient consenting to undergo the study

Exclusion Criteria:

* Indian Race
* Prior treatment for their skin cancer
* More than three synchronous lesions to treatment with RT
* Basal syndrome, xeroderma, vitiligo and albinism
* Immunosuppression
* Prior burn at the tumor site
* Tumor > 5 cm
* Age <18 years
* Carrier mental incapacity
* People in a relationship of dependence as prisoners, soldiers, students, staff, etc..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Rate of complete remission with hypofractionated RT schemes for NMSC. | Second week and twelfth week after initiation of radiotherapy
  RECIST criteria
  * Complete Response: disappearance of the lesion
  * Partial Response: Reduction ≥ 30% of the larger initial diameter of the lesion
  * Progressive Disease: ≥ 20% increase in the largest initial diameter of the lesion
  * Stable disease: not increase enough to consider disease progression or reduction sufficient to consider a partial response.

SECONDARY OUTCOMES:
Quality of Life | Second week and twelfth week after initiation of radiotherapy
  EORTC QLQ-C30
Toxicity | Second week and twelfth week after initiation of radiotherapy
  Late Effects of Normal Tissue (LENT) SOMA Toxicity Grading and Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Nakamura, MD, Principal Investigator — Barretos Cancer Hospital - Fundação Pio XII
Locations (1):
- Barretos Cancer Hospital - Fundacao Pio XII, Barretos, São Paulo, Brazil